CLINICAL TRIAL: NCT04022148
Title: A Nonrandomized, Non-double Blinded Prospective Cohort Study to Evaluate the Preventive Efficacy of Quadrivalent HPV6/11/16/18 Vaccine for the Persistent Infection of HPV16 Genotype or HPV18 Genotype in Japanese Women Aged 27-45 Years.
Brief Title: The Prospective Cohort Study to Evaluate the Preventive Efficacy of HPV Vaccine in Japanese Women Aged 27-45 Years
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Fukui (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Yoshio Yoshida, Professor, University of Fukui
Other Study IDs: C2018001F
Record Dates: First submitted 2019-07-14; First posted 2019-07-16 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Cancer of Cervix; Vaccinia
Keywords: uterine cervical cancer; HPV vaccine; cancer screening
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vaccinia | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Biological: Gardasil — Experimental arm: Vaccine group VS Control arm: Non-Vaccine group

SUMMARY:
A nonrandomized, non-double blinded prospective cohort study to evaluate the preventive efficacy of quadrivalent HPV6/11/16/18 vaccine for the persistent infection of HPV16 genotype or HPV18 genotype in Japanese women aged 27-45 years.

DETAILED DESCRIPTION:
A series of evidence for HPV vaccines has demonstrated the efficacy in young women (Aged less than 26) across the globe. In contrast, limited evidence are available for the efficacy of the quadrivalent HPV6/11/16/18 vaccine in adult women (Aged 27+). Most importantly, evidence for Japanese adult women is not available to date. Nevertheless, , we hypothesize that the quadrivalent HPV6/11/16/18 vaccine demonstrate the efficacy also in Japanese adult women. The outcome from this trial will be the first local evidence, which brings a considerable impact in OB/GY academia where local evidence is weighed heavily compared with global evidence - serves as a strong basis to support catch up program of HPV vaccines for young adults. As a consequence, we believe this study will develop a local supportive evidence for prevention of HPV infection by an HPV vaccine in young adults, which results in substantial public health improvement through prevention of HPV infection in Japan where active recommendation is halted long time.

ELIGIBILITY:
Inclusion Criteria:

* Women with normal cytology results confirmed in cervical cancer screening programs from May 2019 to March 2020
* 27-45 years-old
* Intact uterus
* Willing to undergo the HPV-DNA test (cobas4800) within 12 months

Exclusion Criteria:

* Pregnant women
* Undergo treatment or the follow-up evaluation for CIN within the previous 12 months

  * Previously administered HPV vaccine

Ages: 27 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Japanese adult women (aged 27-45 years) undergo the cervical cancer screening.
Sampling Method: Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of the persistent infection | 48months
  Persistent infection is the cases that the cells from women with HPV16/18 genotype overexpressed p16 and Ki67.

CONTACTS AND LOCATIONS:
Overall Officials: Tetsuji Kurokawa, A, Study Chair — University of Fukui

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kurokawa T, Yamamoto M, Onuma T, Tsuyoshi H, Shinagawa A, Chino Y, Yoshida Y. The study protocol of the evaluation for the preventive efficacy of the HPV vaccine for persistent HPV16/18 infection in Japanese adult women: the HAKUOH study. BMC Cancer. 2020 Nov 3;20(1):1056. doi: 10.1186/s12885-020-07563-0. PMID 33143690